CLINICAL TRIAL: NCT05264662
Title: Pertussis Vaccination Among HIV-infected and HIV-uninfected Pregnant Women
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Farzanah Laher (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Farzanah Laher, Dr, University of Witwatersrand, South Africa
Organization: University of Witwatersrand, South Africa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Maternal Pertussis
Record Dates: First submitted 2022-01-24; First posted 2022-03-03 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: dTap Vaccine
Keywords: Antibodies; Pertussis
MeSH Terms: conditions — Whooping Cough | interventions — adacel

STUDY DESIGN:
Intervention Model Description: open label phase IV clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Open label Adacel (Active Comparator): Tdap (Adacel) ADACEL (0,5 ml) should be administered as an injection by the intramuscular route.
  Re-dosing with ADACEL can be used to boost immunity to diphtheria, tetanus and pertussis at 5- to 10-year intervals.
  ADACEL may be administered to pregnant women during the second and third trimester to provide passive protection to infants against pertussis.
  Interventions: Drug: Adacel (Tdap)
- control (No Intervention): Infants born to unvaccinated mothers.

INTERVENTIONS:
Drug: Adacel (Tdap) — Administer Adacel to hiv infected and hiv uninfected pregnant mothers
  Arms: Open label Adacel

SUMMARY:
Pertussis (also known as whooping cough) is a highly contagious, vaccine-preventable respiratory tract disease, caused by the bacteria Bordetella pertussis. It can affect people of all ages, however young unimmunised or partially immunised infants are the most vulnerable group with the highest rates of complications and death. Recent surveillance data and an increase in the number of pertussis outbreaks being reported nationally, indicate an increase in the incidence of pertussis disease in South Africa.To date there is no data on the effect of vaccinating HIV-infected pregnant women with pertussis-containing vaccines, although there is no reason to think that vaccinating these women would be harmful for them or their foetus. The knowledge gaps on the immunogenicity, safety and VE of pertussis vaccination of HIV-infected pregnant women should be addressed. Adacel which is a registered and licensed vaccine manufactured by Sanofi Pasteur, will be tested in this study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age ≥18 years to <39 years (vaccinated group only).
* Gestational age 20-36 weeks documented by the approximate date of the last menstrual period and corroborated by physical or sonargraphic exam (vaccinated group only).
* Documented to be HIV-infected or HIV-uninfected.
* Good general maternal health.
* Able to understand and comply with planned study procedures.
* Able and willing to provide written informed consent for themselves and infant

Exclusion Criteria:

* Receipt of any live licensed vaccine ≤14 days prior to study initiation.
* Any significant (in the opinion of the site investigator) acute illness.
* Use of anti-cancer systemic chemotherapy or radiation therapy ≤48 weeks of study enrolment or has immunosuppression as a result of an underlying illness or treatment.
* Long term use of glucocorticoids, including oral or parenteral prednisone ≥20 mg/day or equivalent for more than 2 consecutive weeks (or 2 weeks total) ≤12 weeks of study entry, or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) ≤12 weeks before study entry (nasal and topical steroids are allowed).
* Receipt of corticosteroids for preterm labour ≤14 days before study entry.
* Receipt of immunoglobulin or other blood products (with exception of Rho D immune globulin) ≤12 weeks prior to enrolment in this study or is scheduled to receive immunoglobulin or other blood products (with the exception of Rho D immune globulin) during pregnancy or for the first 24 weeks after delivery.
* Receipt of IL2, IFN, GMCSF or other immune mediators ≤12 weeks before enrolment.
* Uncontrolled major psychiatric disorder.
* History of a severe adverse reaction to previous vaccines (vaccinated group only).
* Any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* Pregnancy complications (in the current pregnancy) such as pre-term labour, hypertension (BP >140/90 in the presence of proteinuria or BP >150/100, with or without proteinuria or currently on antihypertensive medication) and pre-eclampsia.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 511 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Concentration of antibodies in pregnant women 1 month after vaccination with Tdap. | 24 months
  To measure antibody responses to all Tdap-IPV antigens (diphtheria, tetanus, PT, FHA, PRN, FIM and polioviruses 1, 2 and 3) in HIV-infected compared with HIV-uninfected pregnant women before and one month after Adacel vaccination.
Concentration of antibodies to all Tdap-IPV and Hexavalent antigens in infants. | 24 months
  To measure antibody responses to all Tdap-IPV and Hexavalent antigens (diphtheria, tetanus, PT, FHA, PRN, FIM, Haemophilus influenzae type-b polyribosyl ribitol phosphate [PRP], polioviruses 1, 2 and 3, and hepatitis B) testing in infants born to mothers who received Adacel during pregnancy and those born to mothers not vaccinated, stratified by maternal HIV status.

SECONDARY OUTCOMES:
Transplacental antibody transfer. | 24 months
  To compare the transplacental antibody transfer ratio of all Tdap-IPV antigens to newborns from HIV-infected mothers and those born to HIV-uninfected mothers vaccinated with Adacel during pregnancy.
Vaccination safety | 24 months
  Number of HIV-infected and HIV-uninfected pregnant women with treatment-related adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Chris Hani Baragwanath Academic Hospital, Johannesburg, GP, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nunes MC, Tamblyn A, Jose L, Ntsimane M, Lerotholi N, Machimana C, Taylor A, Laher F, Madhi SA. Immunogenicity of tetanus, diphtheria and acellular pertussis vaccination among pregnant women living with and without HIV. AIDS. 2023 Dec 1;37(15):2305-2310. doi: 10.1097/QAD.0000000000003731. Epub 2023 Oct 3. PMID 37773052